CLINICAL TRIAL: NCT02268877
Title: A Randomized Prospective Analysis of Time to Diagnosis and Length of Stay of Emergency Department Pelvic Ultrasonography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: United States Naval Medical Center, Portsmouth (U.S. Federal Agency); United States Naval Medical Center, San Diego (U.S. Federal Agency); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 11-1444
Record Dates: First submitted 2014-10-16; First posted 2014-10-20 (Estimated); Results first posted 2017-05-31 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Pregnancy
Keywords: ultrasonography; emergency department
MeSH Terms: conditions — Emergencies | interventions — Ultrasonography

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (2):
- Emergency Medicine Physician Ultrasound (Experimental): Patients will receive an ultrasound performed by a credentialed emergency medicine attending or resident. The ultrasound will be transabdominal, transvaginal, or both. The intervention is the personnel who performs the ultrasound.
  Interventions: Other: Emergency Medicine Physician Ultrasound; Device: Ultrasound
- Radiology Tech Ultrasound (Active Comparator): Patients will receive an ultrasound performed by a credentialed radiology department technician. The ultrasound will be transabdominal, transvaginal, or both. This is standard-of-care.
  Interventions: Device: Ultrasound

INTERVENTIONS:
Other: Emergency Medicine Physician Ultrasound — An ultrasound will be performed by an emergency medicine resident or attending physician
  Arms: Emergency Medicine Physician Ultrasound
Device: Ultrasound — An ultrasound will be performed by a radiology department technician

SUMMARY:
The goal of this project is to compare the efficiency of pelvic ultrasounds performed by emergency medicine residents and attending physicians to the efficiency of pelvic ultrasounds performed by the department of radiology.

DETAILED DESCRIPTION:
This study is a randomized, prospective interventional study of pregnant patients presenting to the emergency department with complaints of pelvic pain and/or vaginal bleeding. This study will be conducted at 4 sites across the United States. Patients who are eligible and consent to participate will be randomized to one of two conditions; 1) a pelvic ultrasound that is performed by a certified emergency department attending or physician, or 2) a pelvic ultrasound that is performed by a certified radiology technician (standard-of-care). The time to diagnosis and emergency department length of stay between the two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* have a positive serum or urine beta-human chorionic gonadotropin (hCG)
* estimated gestational age (EGA) of less than 20 weeks
* complaint of pelvic pain and/or vaginal bleeding

Exclusion Criteria:

* prior known documentation of an intrauterine pregnancy
* estimated gestational age (EGA) of greater than 20 weeks
* peritoneal findings on physical examination
* unstable vital signs as deemed appropriate by the attending physician
* prisoners
* open cervix upon physical examination

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 224 (Actual)
Dates: Start 2013-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Kendall, MD, Principal Investigator — Denver Health and Hospital Authority

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kendall JL, Hoffenberg SR, Smith RS. History of emergency and critical care ultrasound: the evolution of a new imaging paradigm. Crit Care Med. 2007 May;35(5 Suppl):S126-30. doi: 10.1097/01.CCM.0000260623.38982.83. PMID 17446770
- [Result] Durham B, Lane B, Burbridge L, Balasubramaniam S. Pelvic ultrasound performed by emergency physicians for the detection of ectopic pregnancy in complicated first-trimester pregnancies. Ann Emerg Med. 1997 Mar;29(3):338-47. doi: 10.1016/s0196-0644(97)70345-7. PMID 9055772
- [Result] Burgher SW, Tandy TK, Dawdy MR. Transvaginal ultrasonography by emergency physicians decreases patient time in the emergency department. Acad Emerg Med. 1998 Aug;5(8):802-7. doi: 10.1111/j.1553-2712.1998.tb02507.x. PMID 9715242
- [Result] Dart RG. Role of pelvic ultrasonography in evaluation of symptomatic first-trimester pregnancy. Ann Emerg Med. 1999 Mar;33(3):310-20. doi: 10.1016/s0196-0644(99)70368-9. PMID 10036346
- [Result] Tayal VS, Cohen H, Norton HJ. Outcome of patients with an indeterminate emergency department first-trimester pelvic ultrasound to rule out ectopic pregnancy. Acad Emerg Med. 2004 Sep;11(9):912-7. doi: 10.1197/j.aem.2004.03.017. PMID 15347539
- [Result] Blaivas M, Sierzenski P, Plecque D, Lambert M. Do emergency physicians save time when locating a live intrauterine pregnancy with bedside ultrasonography? Acad Emerg Med. 2000 Sep;7(9):988-93. doi: 10.1111/j.1553-2712.2000.tb02088.x. PMID 11043992
- [Result] Shih CH. Effect of emergency physician-performed pelvic sonography on length of stay in the emergency department. Ann Emerg Med. 1997 Mar;29(3):348-51; discussion 352. doi: 10.1016/s0196-0644(97)70346-9. PMID 9055773

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Emergency Medicine Physician Ultrasound | Radiology Tech Ultrasound
Started (122 patients were randomized to this arm.) | 122 | 111 (111 patients were randomized to this arm.)
Completed (118 patients received the intervention) | 118 | 106 (106 patients received the intervention.)
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Emergency Medicine Physician Ultrasound | Radiology Tech Ultrasound | Total
Number analyzed (Participants) | 118 | 106 | 224
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 26 [22 to 31] | 26 [22 to 31] | 26 [22 to 31]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 106 | 224
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 118 | 106 | 224

OUTCOME MEASURES:

1. Primary Outcome: Time to Definitive Diagnosis
Description: The time the patient is placed in room to the time that results of the ultrasound (and/or consultative impression made by radiology or obstetrics and gynecology) are documented in patient chart
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Emergency Medicine Physician Ultrasound | Radiology Tech Ultrasound
Number analyzed (Participants) | 118 | 106
minutes | 87 [40 to 179] | 136 [99 to 169]

2. Primary Outcome: Emergency Department Length-of-Stay
Description: The time the patient is placed in room to the time that the patient is discharged/admitted.
Time Frame: 48 hours
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Emergency Medicine Physician Ultrasound | Radiology Tech Ultrasound
Number analyzed (Participants) | 118 | 106
minutes | 181 [110 to 255] | 201 [171 to 257]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 72 hours after receipt of the intervention.
Description: Ectopic pregnancies and intrauterine fetal demise are expected in the given study population, and have been deemed unrelated to the research intervention by the Principal Investigator.
Arm/Group | Emergency Medicine Physician Ultrasound | Radiology Tech Ultrasound
All-Cause Mortality (participants affected / at risk) | 0/118 | 0/106
Serious Adverse Events (participants affected / at risk) | 2/118 | 2/106
Other Adverse Events (participants affected / at risk) | 4/118 | 2/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emergency Medicine Physician Ultrasound (N=118) | Radiology Tech Ultrasound (N=106)
ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emergency Medicine Physician Ultrasound (N=118) | Radiology Tech Ultrasound (N=106)
intrauterine fetal demise (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 2 (2)

LIMITATIONS AND CAVEATS:
This is not a blinded study. As such the performers may have been biased to complete these procedures more quickly than they would be if the study were not taking place.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No